CLINICAL TRIAL: NCT00959153
Title: Extracorporeal Shock Wave Lithotriptor Indicated for Fragmenting Urinary Stones in the Kidney (Renal Pelvis)
Brief Title: Extracorporeal Shock Wave Lithotriptor Indicated for Fragmenting Urinary Stones in the Kidney
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advance Shockwave Technology GmbH (Industry)
Responsible Party: Hugo Stephan, AST
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G080108
Record Dates: First submitted 2009-08-11; First posted 2009-08-14 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Stones
Keywords: Fragmenting of kidney stones; extracorporeal shockwave lithotripsy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kidney stones (Experimental): Kidney stones
  Interventions: Device: LithoSpace Extracorporeal Shockwave Lithotripter

INTERVENTIONS:
Device: LithoSpace Extracorporeal Shockwave Lithotripter — Shockwave therapy to break up kidney stones

SUMMARY:
A total of 20 subjects presenting with urinary stone(s) in the kidney or ureter will be treated with an extracorporeal shockwave lithotripsy device to fragment the stones. Subjects will be followed for 14 days. If at the 14 day follow-up visit the subject continues to present with a stone size 4 mm or greater will have an option of retreatment or other intervention. If the subject consents to be retreated at this time, this subject will be followed up for another 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solitary Urinary stones in the renal pelvis or renal calyces or ureter
* Presence of one stone greater than 4 mm and less than 12 mm

Exclusion Criteria:

* Urinary tract obstruction, acute or unresolved cholecystitis, cholangitis, pancreatitis or obstruction of the biliary duct system
* Impaction of stone to be treated
* Staghorn stones
* Failed or inadequate lithotripsy procedure within 3 months prior to study
* Coagulation abnormalities or anticoagulation therapy
* Pregnant or females of child-bearing potential General, spinal or epidural anesthesia is contraindicated
* Can not be positioned correctly for fluoroscopic imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
stone fragmentation | 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Metropolitan Lithotriptor Associates, Garden City, New York
  - Allied Urological Services, LLC, New York, New York